CLINICAL TRIAL: NCT05858437
Title: Impact of Propionic Acid on Regulatory T Cell Function in Children With Chronic Kidney Disease
Brief Title: Impact of Propionic Acid on Regulatory T Cell Function in Children With CKD
Acronym: Pro-Kids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Heidelberg (Other); University Hospital, Essen (Other); University Hospital of Cologne (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Benjamin Holle, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EA2/195/22
Record Dates: First submitted 2023-04-25; First posted 2023-05-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sodium propionate

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA Intervention (Experimental): The group which receives the PA as a dietary food supplement. A single capsule contains 500mg of sodiumpropionate, which is taken twice daily for 28 days.
  Interventions: Dietary Supplement: Sodium propionate
- Placebo Intervention (Placebo Comparator): The control-group receives a placebo instead of propionate. The placebo contains maltodextrin and the same amount of sodium chloride as compared to the PA intervention. The placebo is taken twice per day for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium propionate — The patients will be randomized to PA or placebo intervention (2:1 randomization).
  After the intervention of 28 days, we conduct an open-label study phase, where all patients are offered a dietary supplement of PA for overall 12 weeks (8 additional weeks for the intervention group and 12 weeks for the placebo group).
  By doing so we are giving every patient the opportunity to take PA and benefit from the possible positive impact on immunsystem and intestinal barrier function.
  Arms: PA Intervention
Other: Placebo — The patients will be randomized to PA or placebo intervention (2:1 randomization).
  After the intervention of 28 days, we conduct an open-label study phase, where all patients are offered a dietary supplement of PA for overall 12 weeks (8 additional weeks for the intervention group and 12 weeks for the placebo group).
  By doing so we are giving every patient the opportunity to take PA and benefit from the possible positive impact on immunsystem and intestinal barrier function.
  Arms: Placebo Intervention

SUMMARY:
Pro-Kids is a multi-center, double-blind, randomized and placebo-controlled intervention study in children with chronic kidney disease. The investigators address the effect of a dietary food supplementation of propionic acid on the immune system and the function of the intestinal barrier in CKD patients treated with hemodialysis.

DETAILED DESCRIPTION:
Chronic inflammation is a major risk factor of cardiovascular disease progression in CKD, irrespective of confounding comorbidities. Based on current knowledge, microbially-derived metabolites such as short chain fatty acids (SCFA) play an important role in the regulation of chronic inflammatory processes in CKD patients. Children with CKD are known to have reduced serum levels of the SCFA propionic acid (PA), as a consequence of both gut microbial dysbiosis and reduced fiber intake. In animal and human studies the impact of PA on function and abundance of regulatory T cells (Treg) has been demonstrated. Consequently, the investigators aim to normalize the PA serum levels by oral PA food supplementation in hemodialysis patients in order to mitigate chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: > 30kg
* CKD G5 treated with hemodialysis
* Continuous hemodialysis treatment for > 3 months
* Clinical stable condition
* Manifestation of CKD within childhood (<18 years)

Exclusion Criteria:

* Disease or dysfunctions, which disqualifies the patient
* Incapacity of contract or any other circumstances, which prohibit the patient or his legal guardians from understanding setup, meaning and entity of the study
* Acute infections
* Immunosuppressive therapy within the last 12 weeks before the start of the study
* Pre-/pro- or postbiotic or antibiotic therapy within the last 4 weeks before the start of the study
* Planned or unplanned hospitalization within in last 4 weeks before the start of the study or during study
* Malignant diseases
* Pregnancy
* chronic gastrointestinal or hepatic diseases (for example chronic inflammatory bowel disease
* alcohol- or drug abuse
* parallel participation on other interventional trials

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in count of regulatory T-cells from baseline to week 4 | Baseline visit (week 0) in comparison to week 4
  Analysis of Treg counts in whole blood (absolute quantification) and peripheral blood mononuclear cells (PBMC; relative quantification) by flow cytometry.

SECONDARY OUTCOMES:
Propionic acid serum levels and targeted metabolomics | Baseline visit (week 0); Week 2; Week 4; Week 12
  Analysis of PA serum levels and other microbially-derived metabolites by GC-MS and LC-MS
Immune cell phenotyping of peripheral blood mononuclear cells (PBMC) | Baseline visit (week 0); Week 2; Week 4; Week 12
  Patients PBMC will be thawed and immune cells we be analyzed using multicolor flow cytometry and mass cytometry. By using a broad range of different antibodies combined in several panels the investigators will analyse distinct T cell subtypes including markers of activation, but also other immune cells (including B cells, dendritic cells, monocytes, natural killer cells). Data will reported in relation to parent populations (e.g. T heller cells in % of T cells).
T regulatory cell (Treg) suppression assay | Baseline visit (week 0); Week 4
  The suppressive capacity of patients Treg will be analyzed by co-cultivation with conventional, stimulated T cells (Tconv) in different proportions (Treg:Tconv). The proliferation of Tconv will be reported.
Single cell RNA sequencing of immune cells | Baseline visit (week 0); Week 4
  Analysis of the transcriptome of immune cells using cellular indexing of transcriptomes and epitopes (CITEseq)
Intestinal barrier function | Baseline visit (week 0); Week 2; Week 4; Week 12
  Analysis of biomarkers for intestinal barrier function, such as sCD14, zonulin-1 and LPS
Taxonomy of the fecal microbiome | Baseline visit (week 0); Week 4
  The taxonomy of the fecal microbiome will be anayzed using 16S RNA amplicon sequencing.
Cardiovascular Phenotyping | Baseline visit (week 0); Week 2; Week 4; Week 12
  Analysis of heart rate over time.
Cardiovascular Phenotyping | Baseline visit (week 0); Week 2; Week 4; Week 12
  Analysis of blood pressure over time.
Cholesterol levels | Baseline visit (week 0); Week 2; Week 4; Week 12
  Cholesterol levels will be assessed using standard clinical lab values.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Gastroenterology, Nephrology and Metabolic Diseases, Charité-Universitätsmedizin Berlin, Berlin, Germany